CLINICAL TRIAL: NCT05988203
Title: A Randomized, Partially Observer-blind, Dose-escalation, Phase I/II Trial Evaluating the Safety and Immunogenicity of Investigational RNA-based Mpox Vaccine Candidates
Brief Title: A Clinical Study Investigating the Safety and Immune Responses After Immunization With Investigational Monkeypox Vaccines
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: BNT166-01; 1006947 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Monkeypox
Keywords: Prevention of mpox; Monkeypox virus; RNA vaccine; Vaccine; mpox; MPXV; Monkeypox
MeSH Terms: conditions — Mpox, Monkeypox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SSA - BNT166a Dose Level (DL)1 (Experimental): One dose level
  Interventions: Biological: BNT166a
- SSA - BNT166a DL2 (Experimental): One dose level
  Interventions: Biological: BNT166a
- SSA - BNT166a DL3 (Experimental): One dose level
  Interventions: Biological: BNT166a
- SSB - BNT166a DL2 (Experimental): One dose level
  Interventions: Biological: BNT166a
- SSD - BNT166a (Experimental): One dose level based on SSA and SSB data
  Interventions: Biological: BNT166a

INTERVENTIONS:
Biological: BNT166a — Multivalent ribonucleic acid (RNA)-based vaccine for active immunization against monkeypox administered as intramuscular injection.

SUMMARY:
This is a dose-escalation, Phase I/II study evaluating the safety, tolerability, reactogenicity and immunogenicity of the investigational RNA-based multivalent vaccine candidate BNT166a for active immunization against monkeypox (mpox).

This study started with substudy A (SSA) and substudy B (SSB) for which recruitment has been completed. A Substudy C (SSC) was planned, but the sponsor decided not to conduct it. This study will therefore continue with substudy D (SSD).

In SSA and SSB, dosing started with an initial sentinel group, followed by the expansion cohort.

This study was initially planned to investigate two vaccine candidates (the quadrivalent BNT166a and the trivalent BNT166c). The sponsor decided to not activate the groups with BNT166c.

DETAILED DESCRIPTION:
Substudy A is an open-label, dose-escalation, Phase I substudy to assess the reactogenicity, safety, and immunogenicity of up to three dose levels of the multivalent vaccine candidate BNT166a in 48 healthy participants with no prior history of known or suspected smallpox vaccination (vaccinia-naïve participants).

Substudy B is a one group, open-label, Phase I substudy to assess the reactogenicity, safety and immunogenicity of the multivalent vaccine candidate BNT166a in 16 healthy participants with prior history of smallpox vaccination (vaccinia-experienced).

Substudy D is a one group, open-label, Phase IIa substudy to assess the reactogenicity, safety, and immunogenicity of one dose level of BNT166a in ~32 healthy participants with no prior history of known or suspected smallpox vaccination (i.e., vaccinia-naïve participants). SSD will be initiated after the interim analysis of SSA and SSB safety, reactogenicity, and immunogenicity data.

The duration of study participation is ~ 14 months per participant in all of the substudies.

ELIGIBILITY:
Inclusion Criteria (applicable to all substudies unless otherwise specified):

* Have given informed consent by signing and dating the informed consent form (ICF) before initiation of any study-specific procedures.
* Are willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study, including the prohibited concomitant medications. This includes that they are able to understand and follow study-related instructions.
* SSA and SSD only: Are 18 through 45 years of age (inclusive) at the time of informed consent.
* SSB only: Are 50 through 65 years of age (inclusive) at the time of informed consent.
* Have a body mass index over 18.5 kg/m^2 and under 30 kg/m^2 and weigh at least 50 kg at Visit 0.
* Are healthy, in the clinical judgment of the investigator based on volunteer-reported medical history data, physical examination, 12-lead electrocardiogram (ECG), vital signs, and clinical laboratory test results.
* SSA and SSD only: Have no prior history of known or suspected smallpox vaccination and no detectable smallpox vaccination characteristic scar (vaccinia-naïve participants).
* SSB only: Have a history of prior smallpox vaccination (i.e., are vaccinia-experienced), determined based on medical records and/or presence of smallpox vaccination characteristic scar. The most recent smallpox vaccination should have been received before 1980.
* Agree not to enroll in another study with an investigational medicinal product starting from Visit 0 and until the end of this study.
* Negative human immunodeficiency virus (HIV)-1 and HIV-2 antigen/antibody blood test result at Visit 0.
* Negative Hepatitis B surface antigen and negative core antibodies test results and negative anti Hepatitis C virus antibodies (anti-HCV), or negative Hepatitis C virus (HCV) polymerase chain reaction test result if the anti-HCV is positive at Visit 0.
* Volunteers of childbearing potential (VOCBP) must not be pregnant. VOCBP and men who are sexually active with partners of childbearing potential and their sexual partners born female should use a highly effective form of contraception from at least 28 days prior to Dose 1 up to at least 90 days after receiving the last dose of study treatment, and should agree not to donate eggs (ova, oocytes) or sperm.

Exclusion Criteria (applicable to all substudies unless otherwise specified):

* History of mpox, smallpox or vaccinia infection based on volunteer-reported medical history.
* Pregnant, breastfeeding, planning pregnancy or planning to father children starting from Visit 0 and continuously until 90 days after receiving Dose 2.
* History of known or suspected severe adverse reaction including allergic reaction (e.g., anaphylaxis) to vaccines or to vaccine components such as lipids.
* Current or history of the following medical conditions at Visit 0 or Visit 1:

  * Uncontrolled, moderate or severe asthma; asthma severity as defined in the US National Asthma Education and Prevention Program Expert Panel report
  * Chronic obstructive pulmonary disease.
  * Diabetes mellitus type 1 or type 2, including cases controlled with diet alone (Not excluded: history of isolated gestational diabetes).
  * Hypertension: If a person has hypertension, exclude for blood pressure that is not well controlled. Well controlled blood pressure is defined as consistently ≤140 mm Hg systolic and ≤90 mm Hg diastolic, with or without medication, with only isolated, brief instances of higher readings, which must be <150 mm Hg systolic and <100 mm Hg.
  * Systolic blood pressure ≥150 mm Hg or diastolic blood pressure ≥100 mm Hg.
  * Malignancy, excluding localized basal or squamous cell cancer.
  * Cardiovascular diseases, (e.g., myocarditis, pericarditis, coronary heart disease, myocardial infarction, congestive heart failure, cardiomyopathy or clinically significant arrhythmias, stroke or transient ischemic attack).
  * Bleeding disorders (e.g., factor deficiency, coagulopathy, or platelet disorder).
  * Seizure disorder: History of seizure(s) within past 3 years; use of medications in order to prevent or treat seizure(s) at any time within the past 3 years.
  * Estimated glomerular filtration rate <60 mL/min/1.73 m^2.
  * Chronic liver disease.
* Schizophrenia, major depressive disorder, suicidal ideation. Such psychiatric illnesses, as bipolar disorder, autism and attention deficit-hyperactivity disorder that at the discretion of the investigator could interfere with participation and follow-up as outlined by the study.
* Current or history of the following diseases associated with immune dysregulation:

  * Known or suspected immunodeficiency.
  * History of solid organ or bone marrow transplantation.
  * Asplenia: any condition resulting in the absence of a functional spleen.
  * Currently existing or history of any autoimmune disease.
* SSA and SSB: At Visit 0, any screening hematology and/or blood chemistry laboratory value that meets the definition of a Grade ≥1 abnormality (according to the FDA toxicity grading scale; see separate exclusion criteria for bilirubin and troponin I). Individuals with any stable Grade 1 abnormalities may be considered eligible at the discretion of the investigator. A stable Grade 1 laboratory abnormality is defined as the value which is ≤ Grade 1 upon repeated testing on a second sample from this individual during the screening period (prior to Visit 1). Individuals with abnormal but not clinically significant parameters not included in the FDA toxicity guidance may be considered eligible at discretion of investigator.
* SSD only: At Visit 0, any screening hematology and/or blood chemistry laboratory value (according to the FDA toxicity grading scale) that meets the definition of a Grade ≥2 abnormality; individuals with clinically non-significant Grade 1 abnormalities may be considered eligible at the discretion of the investigator. Individuals with abnormal but clinically non-significant parameters not included in the FDA toxicity guidance may be considered eligible at the discretion of the investigator. See separate exclusion criteria for bilirubin and troponin I.
* Abnormal total bilirubin at Visit 0. Note: inclusion of volunteers with bilirubin ≤1.25 upper limit of normal (ULN) if due to Gilbert's syndrome is allowed.
* Any abnormal troponin I value at Visit 0.
* A 12-lead ECG at Visit 0 which is consistent with probable or possible myocarditis/pericarditis or which demonstrates clinically relevant abnormalities that may affect participant safety or are otherwise clinically significant findings (e.g., complete left bundle branch block, AV block, average corrected QT interval by Fridericia (QTcF interval) >450 msec, signs of myocardial infarction, ST elevation consistent with myocardial ischemia, or serious brady- or tachyarrhythmias).
* Febrile illness (body temperature ≥38.0°C) or other acute illness within 48 hours prior to Dose 1 and/or current (if presented at Visit 1, temporary deferral is allowed).
* Participation or planned participation in strenuous or endurance exercise within 7 days before or after each IMP administration.
* SSA and SSD only: Vaccination with any Orthopoxvirus-based vaccine including vaccines for prevention of smallpox, disease caused by vaccinia virus or mpox, or vector Orthopoxvirus-based vaccines.
* SSB only: Vaccination for prevention of mpox or disease caused by vaccinia virus, or with vector Orthopoxvirus-based vaccine. Vaccination for prevention of smallpox done in or after 1980.
* Any vaccination within 28 days before Dose 1. Seasonal inactivated influenza vaccine is allowed, however, it should be administered at least 14 days before IMP administration.
* Any non-study IMP within 28 days or five half-lives (whichever is longer) before Dose 1.
* Blood/plasma products and/or immunoglobulins within 120 days before Dose 1.
* Allergy treatment with antigen injections within 14 days before Dose 1.
* Immunosuppressive therapy, including corticosteroids, or radiotherapy within 6 months or five half-lives (whichever is longer) before Dose 1. If systemic corticosteroids have been administered short term (≤14 days, at a dose of ≤20 mg/day of prednisone or equivalent) for treatment of an acute illness, individuals should be enrolled in the study only after corticosteroid therapy has been discontinued for at least 28 days before Dose 1. Intraarticular, intrabursal, or topical (skin or eyes) corticosteroids are permitted.
* Have a history of alcohol abuse within 1 year before Visit 0 or have a history of substance abuse within the past 5 years before Visit 0.
* Are vulnerable individuals as per ICH E6 definition, i.e., are individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
SSA, SSB, and SSD - Proportion (%) of participants reporting solicited local reactions at the injection site (pain, erythema/redness, induration/swelling) | From Dose 1 through Day 7 post-Dose1 inclusive; and from Dose 2 through Day 7 post-Dose 2 inclusive
  For each group
SSA, SSB, and SSD - Proportion (%) of participants reporting solicited systemic events (vomiting, diarrhea, headache, fatigue, myalgia, arthralgia, chills, and fever) | From Dose 1 through Day 7 post-Dose1 inclusive; and from Dose 2 through Day 7 post-Dose 2 inclusive
  For each group
SSA, SSB, and SSD - Proportion (%) of participants with at least one unsolicited adverse event (AE) occurring from Dose 1 through Day 28 post-Dose 1 inclusive | From Dose 1 through Day 28 post-Dose 1 inclusive
  For each group
SSA, SSB, and SSD - Proportion (%) of participants with at least one unsolicited AE occurring from Dose 2 through Day 28 post-Dose 2 inclusive | from Dose 2 through Day 28 post-Dose 2 inclusive
  For each group
SSA, SSB, and SSD - Proportion (%) of participants with at least one serious adverse event (SAE) occurring from Dose 1 through Day 201 post-Dose 1 inclusive | From Dose 1 through Day 201 post-Dose 1 inclusive
  For each group
SSA, SSB, and SSD - Proportion (%) of participants with at least one adverse event of special interest (AESI) occurring from Dose 1 through Day 201 post-Dose 1 inclusive | From Dose 1 through Day 201 post-Dose 1 inclusive
  For each group

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (8):
- United States (4):
  - California Research Foundation, San Diego, California
  - Alliance for Multispecialty Research, LLC, Kansas City, Missouri
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - University of Washington Virology Research Clinic, Seattle, Washington
- United Kingdom (4):
  - Addenbrooke's Hospital - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Royal Surrey County Hospital Foundation Trust, NIHR Royal Surrey Clinical Research Facility, Guildford
  - Guy's and St Thomas' NHS Foundation Trust of St Thomas' Hospital, London
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuiani A, Dulberger CL, De Silva NS, Marquette M, Lu YJ, Palowitch GM, Dokic A, Sanchez-Velazquez R, Schlatterer K, Sarkar S, Kar S, Chawla B, Galeev A, Lindemann C, Rothenberg DA, Diao H, Walls AC, Addona TA, Mensa F, Vogel AB, Stuart LM, van der Most R, Srouji JR, Tureci O, Gaynor RB, Sahin U, Poran A. A multivalent mRNA monkeypox virus vaccine (BNT166) protects mice and macaques from orthopoxvirus disease. Cell. 2024 Mar 14;187(6):1363-1373.e12. doi: 10.1016/j.cell.2024.01.017. Epub 2024 Feb 15. PMID 38366591